CLINICAL TRIAL: NCT04325425
Title: Folfirinox Versus Platinum - Etoposide as First Line Chemotherapy for Metastatic Grade 3 Poorly Differentiated Neuroendocrine Carcinoma of Gastro Entero Pancreatic and Unknown Primary Associated With Molecular Profiling for Therapeutic Targets & Predictive Biomarkers Identification
Brief Title: Chemotherapy For Metastatic Grade 3 Poorly Differentiated NEuroendocrine Carcinoma Of GastroEnteroPancreatic And Unknown Primary
Acronym: FOLFIRINEC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE 69
Record Dates: First submitted 2020-02-25; First posted 2020-03-27 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Neuroendocrine Carcinoma
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — FOLFOXIRI protocol; Cisplatin; Carboplatin

STUDY DESIGN:
Intervention Model Description: mFOLFIRINOX (experimental arm) vs Platinum - Etoposide (standard arm)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mFOLFIRINOX (Experimental): mFOLFIRINOX will be administered once every 14 days for up to 12 cycles. One cycle consists of 14 days (2 weeks) with injection on D1 of each cycle (D1=D15). Patients are eligible for repeated treatment cycles in the absence of disease progression and undue adverse events.
  Interventions: Drug: FOLFOXIRI Protocol
- platinum - etoposide (Active Comparator): Platinum-Etoposide regimen will be administered once every 21 days. Treatment will be continued for 6 to 8 cycles or 24 weeks maximum. One cycle consists of 21 days (3 weeks) with injection on D1 of each cycle (D1=D22). Patients are eligible for repeated treatment cycles in the absence of disease progression and undue adverse events.
  Interventions: Drug: Cisplatin injection

INTERVENTIONS:
Drug: FOLFOXIRI Protocol — Platinum-Etoposide regimen will be administered once every 21 days. Treatment will be continued for 6 to 8 cycles or 24 weeks maximum. One cycle consists of 21 days (3 weeks) with injection on D1 of each cycle (D1=D22). Patients are eligible for repeated treatment cycles in the absence of disease progression and undue adverse events.
  Other Names: modified FOLFIRINOX
  Arms: mFOLFIRINOX
Drug: Cisplatin injection — Cisplatin 100 mg/m2, IV infusion over 3 hours or Carboplatin AUC 5, IV infusion over 30 minutes on day 1 [the dose of carboplatin will be determined for each cycle using the Calvert's formula (carboplatin dose (mg) = target AUC 5 x estimated glomerular filtration rate (eGFR, mL/min) + 25)];
  • Etoposide 100 mg/m² IV infusion over 1 hour on day 1,2 and 3
  Other Names: Platinum - Etoposide; carboplatin injection
  Arms: platinum - etoposide

SUMMARY:
there is a need for improving chemotherapy regimen for metastatic G3 NEC of GEP and Unknown origin and this goal may be achieved through more "personalized" chemotherapy regimen.the hypothesis is that mFOLFIRINOX regimen could be a good candidate for challenging the platinum-etoposide regimen in patients with metastatic G3 NEC of GEP or unknown origin. Furthermore, in order to get insights in the putative predictive biomarkers of efficacy of these two regimens, an effort toward a precise molecular characterization of these tumors is required in order to be able to define which subgroup of G3 NEC needs to be treated by which chemotherapy regimen. The FOLFIRINEC trial is set up in order to try to answer these questions

DETAILED DESCRIPTION:
Grade 3 poorly differentiated neuroendocrine carcinomas (G3 NEC) are rare diseases. The diagnosis is often done at the metastatic stage and the prognosis is poor. The standard first-line treatment is the platinum-etoposide chemotherapy regimen, mostly based on retrospective studies .With this regimen, response rate (RR) is 40 to 70% but the median progression-free survival is between 4 and 9 months. Disease progression almost always occurs during or just after treatment and median overall survival (OS) is only about 12-15 months for gastro-entero-pancreatic (GEP) NEC with similar efficacy of either cisplatin or carboplatin in the NORDIC study and of 8 to 10 months for pulmonary NEC. After progression, only 40 to 45% of patients will receive a second line chemotherapy which will include 5-fluoro-uracil (5FU) and irinotecan (FOLFIRI or oxaliplatin (XELOX, FOLFOX).This second line treatment can provide around 30% of responses and a median progression-free survival of 4 months. Taken together, these data indicate a major medical need for improving G3 NEC treatments.

Few trials have tried to challenge the standard platinum-etoposide first-line treatment. Clinical trials challenging the platinum-etoposide combination in the first-line setting feasibility has already been demonstrated with paclitaxel-carboplatin-etoposide combination and the cisplatin-irinotecan phase III trials. However, these trials have shown equivalent activities between experimental group and platinum-etoposide regimen. Furthermore, the lack of randomization precluded any definitive conclusion. Therefore, prospective randomized studies aiming at improving first-line chemotherapy remains challenging and clinically meaningful. Currently, the only randomized trial in progress in first line treatment of metastatic G3 GEP NEC compares platinum-etoposide to temozolomide-capecitabine. Other mono-arm phase II studies evaluate carboplatin - nab-paclitaxel and everolimus - temozolomide combinations. FOLFIRINOX is also planned to be evaluated in a mono-arm first or subsequent line setting at Lee. H Moffit Cancer Institute.

Although the second-line treatment studies of metastatic G3 NEC of GEP or unknown origin were retrospective, they have suggested that both irinotecan and oxaliplatin, in conjunction with 5FU can have anti-tumor effect in G3 NEC. In recent years, the intensified chemotherapy regimen FOLFIRINOX, which associates 5FU, oxaliplatin and irinotecan, has shown great efficacy in several digestive cancer such as pancreas or colorectal adenocarcinoma. Tolerance of this regimen has improved over the years with better management and dose adaptations that has led to the development of the mFOLFIRINOX regimen . mFOLFIRINOX could be a good first-line treatment candidate in metastatic GEP NEC because: (i) Oxaliplatin, irinotecan and 5FU have anti tumor effect in metastatic GEP NEC; (ii) trichemotherapy with a potential high RR could be efficient in these chemosensitive cancers; (iii) the degradation of performance status following tumor progression after first-line treatment makes access to a second line uncertain which argue for the use of an aggressive first-line treatment; (iiii) administration on a one-day outpatient basis (day hospital) as well as acceptable and manageable side effects, could have an impact on quality of life in these patients with a poor prognosis. the hypothesis is that the intensive trichemotherapy mFOLFIRINOX, improves the prognosis of patients with metastatic G3 NEC from GEP or unknown primary.

Little is known on the predictive factors of first-line chemotherapy in metastatic G3 NEC and few trials have tried to challenge the platinum-etoposide standard. Among G3 NEC, there are 2 histological subtypes; eg. small cell NEC (SCNEC) and large cell NEC (LCNEC). These two subtypes are treated with the same platinum-etoposide regimen, whatever the primary, although RR seem to differ between SCNEC and LCNEC. This difference has been reported for pulmonary G3 NEC: the RR to platinum-etoposide was 34% in the French phase II trial on LCNEC and 37% in a recent retrospective study, while the RR of SCNEC was 50 to 60% in different reports. Moreover, the difference in RR to platinum based chemotherapy has also been recently reported in a Japanese retrospective study of pancreatic NEC with RR of 68 and 44% for SCNEC and LCNEC respectively.

These results suggest that there could be some biological differences among G3 NEC, which could be responsible for the different responses to treatment and that G3 NEC could be a heterogeneous group of tumors. While pulmonary SCNEC are fairly homogeneous tumors and are characterized by a quasi-constant Rb loss of expression, LCNEC are more heterogeneous. A sequencing study of 45 pulmonary LCNEC samples has shown that 40% of the tumors had a mutational profile which looks like small cell lung cancer (SCLC) while 58% of the tumors had a mutation profile like those found in non-small cell lung cancer (NSCLC) (Rekhtman et al. 2016). According to their molecular profiles, LCNEC could be divided between "NSCLC-like" and "SCLC-like" tumors. "SCLC-like" tumors were characterized by p53 and Rb inactivating mutations while "NSCLC-like" tumors were characterized by p53 inactivating mutations but also KRAS and STK11 mutations like those found in lung adenocarcinomas. Therefore, when considering the pulmonary NEC model, it could be hypothesized that, among LCNEC, some tumors may be "adenocarcinoma-like" and some other may be really "SCNEC-like". This hypothesis is supported by some data from digestive tract G3 NEC. Rb loss of expression is found in 100% of SCNEC of the colon versus 31% of LCNEC of the colon; Rb loss is also found in 89% of SCNEC versus 60% of LCNEC of the pancreas . These data seem to parallel the pulmonary NEC data and suggest that G3 NEC, especially LCNEC, is a heterogeneous group of tumors with some of them being biologically very close to SCNEC with Rb loss and others being more biologically close to adenocarcinoma. G3 SCNEC are probably more homogeneous but some heterogeneity is also possible within this group because the pathological diagnosis of "large"versus "small cell" is challenging. This has led to the hypothesis that LCNEC could arise from different cell of origin, i.e; from neuroendocrine precursors and/or from trans-differentiation of adenocarcinoma cells as already described in prostate and lung cancer while SCNEC would represent the bona fide poorly differentiated NEC.

Taking together the putative biological heterogeneity of G3 NEC and the need, in clinical practice, for more effective chemotherapy regimen, it can be hypothesized that a more "tailored" chemotherapy regimen is needed for G3 NEC patients. This is supported by the retrospective analysis from the Dutch registry of pulmonary NEC which have suggested that "NSCLC-like" chemotherapy regimen without pemetrexed were more effective than "SCLC-like" chemotherapy regimen for the treatment of pulmonary LCNEC. Moreover, the same group has recently reported that the better efficacy of "NSCLC-like" chemotherapy was observed for pulmonary LCNEC without Rb mutation (the so-called "NSCLC-like" tumors in the Rekhtman et al study) while Rb mutated LCNEC did not have significantly different response to "SCLC-like" and "NSCLC like" chemotherapy regimens. This has also been shown in pancreatic LCNEC with a RR to first-line platinum-based chemotherapy of 80% in case of Rb loss of expression, and 38.4% in case of retained Rb expression.

ELIGIBILITY:
Inclusion Criteria:

* Grade 3 neuroendocrine carcinoma or high grade MiNEN with a grade 3 poorly differentiated neuroendocrine carcinoma component ≥30% of gastro-entero-pancreatic or unknown primary

  * Poorly differentiated
  * Small cell or large cell or non-small cell or non- typeable
  * Metastatic disease
  * First-line, no prior therapy for metastatic disease, no prior use of carboplatin, oxaliplatin, cisplatin, etoposide, irinotecan and 5-fluorouracile
  * At least one measurable lesion as assessed by CT-scan or MRI according to RECIST 1.1 guidelines
  * Available tumor block
  * ANC ≥ 1.5x109/l, platelet ≥ 100x109/l and hemoglobin > 8 g/dl
  * Total bilirubin ≤ 1.5N, AST ≤ 2.5N, ALT≤ 2.5N or AST/ALT ≤ 5N in case of liver metastases.
  * Age ≥ 18 years
  * ECOG Performance Status ≤ 1
  * Signed and dated informed consent, and willing and able to comply with protocol requirements.
  * Women of childbearing potential, as well as men (who have sexual relations with women of childbearing potential) must agree to use an effective method of contraception throughout this study and during the 15 months following administration of the last dose of the study medicinal product
  * Patient who is a beneficiary of the Social security system

Exclusion Criteria:

* Grade 3 well differentiated neuroendocrine tumor according to WHO 2017 classification

  * Severe renal impairment (creatinine clearance less than 30 mL/min, MDRD)
  * Partial or complete Dihydropyrimidine Dehydrogenase (DPD) deficiency (uracilemia ≥ 16 ng/mL)
  * Gilbert's syndrome
  * Pre-existing permanent neuropathy (NCI CTC V4.0 grade ≥2)
  * Previously treated by chemotherapy or targeted therapy
  * Brain metastases unless they are asymptomatic or under stable corticosteroid doses for 2 weeks otherwise. Radiation therapy prior to inclusion is required if symptomatic.
  * Combination with sorivudine and others analogues as brivudine (irreversibly inhibits the enzyme dihydropyrimidine dehydrogenase)
  * Treatment with St John's Wort (Hypericum perforatum)
  * Pregnant women or breastfeeding mother
  * Known or historical active infection with HIV, or known active infection untreated with hepatitis B or hepatitis C
  * History of prior malignancy, except for cured non-melanoma skin cancer, cured in situ cervical carcinoma, or other treated malignancies with no evidence of disease for at least three years.
  * Active or suspected acute or chronic uncontrolled disease that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study
  * vaccinations (live vaccine) within 30 days prior to start of study drugs
  * Patient under guardianship and/or deprived of his/her freedom
  * QT/QTc interval > 450 msec for male and > 470 msec for female at EKC.
  * K+ < LLN, Mg²+ < LLN, Ca²+ < LLN
  * History or know hypersensitivity to any of the study chemotherapy agents, or their excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
median of progression free survival | 7.5 MONTHS
  The primary endpoint is the median of progression-free survival. PFS is defined as the time interval between date of randomization and date of the first radiological progression (according to RECIST 1.1) or death due to any cause, whichever occurs first, according to investigator. Patient alive without progression will be censored at date of last follow-up visit.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 9 MONTHS
  time interval between date of randomization and date of the first radiological progression (according to RECIST 1.1) or death due to any cause, whichever occurs first, according to the centralized review.
Overall survival | 15 MONTHS
  OS is defined as the time interval between date of randomization and date of death (whatever the cause). Patients alive will be censored at date of last news.
Best objective response rate | 8 weeks after randomization
  The best objective response rate is defined as the proportion of patients with an objective response (Complete response (CR) + Partial response (PR)) at any evaluation during the treatment, according to RECIST 1.1.
Safety and tolerability profile: percentage of patients who experienced toxicities | 24 months after randomization of the last subject
  Safety profile is defined as the percentage of patients who experienced toxicities and grading of these toxicities. Toxicities will be presented as the number of patients presenting at least an episode of toxicity by maximum grade. Toxicity grading will follow NCI-CTC V4 guidelines

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Chu de Caen, Caen
  - Chu Dijon Bourgogne, Dijon
  - Institut de Cancérologie de Bourgogne, Dijon
  - Chu de Limoges - Dupuytren, Limoges
  - Centre Hospitalier de Saint Malo, St-Malo
  - CH de Troyes, Troyes

IPD SHARING:
Plan to Share IPD: Undecided